CLINICAL TRIAL: NCT03178552
Title: A Phase II/III Multicenter Study Evaluating the Efficacy and Safety of Multiple Targeted Therapies as Treatments for Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) Harboring Actionable Somatic Mutations Detected in Blood (B-FAST: Blood-First Assay Screening Trial)
Brief Title: A Study to Evaluate the Efficacy and Safety of Multiple Targeted Therapies as Treatments for Participants With Non-Small Cell Lung Cancer (NSCLC)
Acronym: B-FAST
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29554; 2017-000076-28 (EudraCT Number)
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; atezolizumab; Pemetrexed; Cisplatin; Carboplatin; Gemcitabine; entrectinib; cobimetinib; Vemurafenib; Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort A: Alectinib 600 Milligrams (mg) (Experimental): This cohort includes participants with anaplastic lymphoma kinase (ALK) positive NSCLC. Participants will receive alectinib 600 mg orally twice in a day (BID) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Enrollment to Cohort A is complete.
  Interventions: Drug: Alectinib
- Cohort B: Dose Finding Phase (DFP) Alectinib (Experimental): This cohort includes participants with rearranged during transfection (RET) positive NSCLC. Participants may receive alectinib 900 or 1200 mg orally BID until disease progression, unacceptable toxicity, withdrawal of consent or death if the recommended phase 2 dose (RP2D) is not established in any other clinical study. Participants may receive 750 mg or 600 mg, if it is unsafe to pursue the higher starting dose.
  Enrollment to Cohort B is complete.
  Interventions: Drug: Alectinib
- Cohort B: Dose Expansion Phase (DEP) Alectinib (Experimental): This cohort includes participants with RET positive NSCLC. Participants will receive alectinib at the RP2D established in the DFP of Cohort B or a separate clinical study. Participants will continue receiving study treatment until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Enrollment to Cohort B is complete.
  Interventions: Drug: Alectinib
- Cohort C: Atezolizumab 1200 mg (Experimental): This cohort includes participants with bTMB positive NSCLC. Participants will receive atezolizumab at a dose of 1200 mg administered by IV infusion every 21 days (Q21D) until disease progression, loss of clinical benefit, unacceptable toxicity, withdrawal of consent or death.
  Enrollment to Cohort C is complete.
  Interventions: Drug: Atezolizumab
- Cohort C: Pemetrexed, Cisplatin or Carboplatin (Active Comparator): This cohort includes participants with bTMB positive, non-squamous NSCLC. Participants will receive 4 or 6 cycles of treatment, with each cycle being 21 days in duration. Carboplatin at a dose of area under the concentration-time curve (AUC) of 5 or 6 IV or cisplatin at a dose of 75 milligrams per meter square (mg/m^2) IV on Day 1 of each cycle combined with pemetrexed at a dose of 500 mg/m^2 IV on Day 1 of each cycle. Pemetrexed may be continued as maintenance therapy every 21 days (Q21D) as per local standard of care.
  Enrollment to Cohort C is complete.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Cohort C: Gemcitabine, Cisplatin or Carboplatin (Active Comparator): This cohort includes participants with bTMB positive, squamous NSCLC. Participants will receive 4 or 6 cycles of treatment, with each cycle being 21 days in duration. Gemcitabine 1250 mg/m^2 IV on Days 1 and 8 of every cycle and cisplatin 75 mg/m^2 IV on Day 1 Q21D or gemcitabine 1000 mg/m^2 IV on Days 1 and 8 of every cycle and carboplatin AUC 5 IV on Day 1 Q21D.
  Enrollment to Cohort C is complete.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine
- Cohort D: Entrectinib 600 Milligrams (mg) (Experimental): This cohort includes participants with c-ros oncogene 1 positive (ROS1+) NSCLC. Participants will receive entrectinib 600 mg orally once a day (QD) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Enrollment to Cohort D is complete.
  Interventions: Drug: Entrectinib
- Cohort E: Atezolizumab, Vemurafenib, and Cobimetinib (Experimental): This cohort includes participants with BRAF V600 mutation. Participants will receive: atezolizumab 1680 mg IV Q4W after the run-in period; cobimetinib 60 mg orally (PO) QD on Days 1-21 of each cycle during the run-in and triple-combination periods; and vemurafenib 960 mg PO twice daily (BID) on Days 1-21 of the initial run-in period, then 720 mg PO BID on Days 1-22 of the initial run-in period and on Days 1-28 of each cycle during the triple-combination period.
  Enrollment to Cohort E is complete.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib; Drug: Vemurafenib
- Cohort F: Atezolizumab, Bevacizumab, Carboplatin, and Pemetrexed (Experimental): This cohort includes participants with EGFR exon 20+ NSCLC. Participants will receive atezolizumab + bevacizumab + carboplatin + pemetrexed for 4 or 6 induction cycles (cycle = 21 days). After induction therapy, participants will continue maintenance treatment with atezolizumab + bevacizumab + pemetrexed until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Enrollment to Cohort F is complete.
  Interventions: Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Bevacizumab
- Cohort G: Divarasib or Docetaxel (Experimental): Experimental: Cohort G: GDC-6036 or Docetaxel This cohort includes participants with KRAS G12C mutation. Participants will receive GDC-6036 PO QD or IV docetaxel Q3W (75 mg/m^2) until disease progression or unacceptable toxicity
  New participants will no longer receive docetaxel.
  Interventions: Drug: Divarasib; Drug: Docetaxel
- Cohort Z: Natural History Cohort (No Intervention): Participants with genomic profiles of interest that are not enrolled in the other cohorts will enter into natural history follow-up.

INTERVENTIONS:
Drug: Alectinib — Participants will receive 600 mg BID (Cohort A); 900, 1200, or 750 mg BID (Cohort B) or RP2D BID; orally until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Other Names: RO5424802
  Arms: Cohort A: Alectinib 600 Milligrams (mg); Cohort B: Dose Expansion Phase (DEP) Alectinib; Cohort B: Dose Finding Phase (DFP) Alectinib
Drug: Atezolizumab — Participants will receive atezolizumab 1200 mg IV infusion Q21D (Cohorts C and F) or 1680 mg IV infusion Q4W starting on Day 29 (Cohort E).
  Other Names: RO5541267
  Arms: Cohort C: Atezolizumab 1200 mg; Cohort E: Atezolizumab, Vemurafenib, and Cobimetinib; Cohort F: Atezolizumab, Bevacizumab, Carboplatin, and Pemetrexed
Drug: Pemetrexed — Participants will receive pemetrexed 500 mg/m^2 IV infusion on Day 1 Q21D.
  Arms: Cohort C: Pemetrexed, Cisplatin or Carboplatin; Cohort F: Atezolizumab, Bevacizumab, Carboplatin, and Pemetrexed
Drug: Cisplatin — Participants will receive cisplatin 75 mg/m^2 IV on Day 1 Q21D.
  Arms: Cohort C: Gemcitabine, Cisplatin or Carboplatin; Cohort C: Pemetrexed, Cisplatin or Carboplatin
Drug: Carboplatin — Participants will receive carboplatin of AUC 5 or 6 IV on Day 1 Q21D.
  Arms: Cohort C: Gemcitabine, Cisplatin or Carboplatin; Cohort C: Pemetrexed, Cisplatin or Carboplatin; Cohort F: Atezolizumab, Bevacizumab, Carboplatin, and Pemetrexed
Drug: Gemcitabine — Participants will receive gemcitabine 1000 or 1250 mg/m^2 on Days 1 and 8 of every cycle (1 Cycle=21 days).
  Arms: Cohort C: Gemcitabine, Cisplatin or Carboplatin
Drug: Entrectinib — Participants will receive entrectinib 600 mg orally QD.
  Other Names: RO7102122
  Arms: Cohort D: Entrectinib 600 Milligrams (mg)
Drug: Cobimetinib — Participants will receive 60 mg PO QD on Days 1-21 of the initial run-in and triple-combination periods.
  Other Names: RO5514041
  Arms: Cohort E: Atezolizumab, Vemurafenib, and Cobimetinib
Drug: Vemurafenib — Participants will receive 960 mg PO BID on Days 1-21 of the initial run-in period, and 720 mg PO BID on Days 22-28 of the initial run-in period and on Days 1-28 of each cycle during the triple-combination period.
  Other Names: RO5185426
  Arms: Cohort E: Atezolizumab, Vemurafenib, and Cobimetinib
Drug: Bevacizumab — Participants will receive 15 mg/kg of IV bevacizumab on Day 1 of each 21-day cycle during the induction and maintenance periods.
  Other Names: RO4876646
  Arms: Cohort F: Atezolizumab, Bevacizumab, Carboplatin, and Pemetrexed
Drug: Divarasib — Participants will receive divarasib PO QD until disease progression or unacceptable toxicity.
  Other Names: RO7435846; GDC-6036
  Arms: Cohort G: Divarasib or Docetaxel
Drug: Docetaxel — Participants will receive IV docetaxel Q3W (75 mg/m^2) until disease progression or unacceptable toxicity
  Arms: Cohort G: Divarasib or Docetaxel

SUMMARY:
This is a phase 2/3, global, multicenter, open-label, multi-cohort study designed to evaluate the safety and efficacy of targeted therapies or immunotherapy as single agents or in combination in participants with unresectable, advanced or metastatic NSCLC determined to harbor oncogenic somatic mutations or positive by tumor mutational burden (TMB) assay as identified by a blood-based next-generation sequencing (NGS) circulating tumor DNA (ctDNA) assay.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of unresectable Stage IIIb not amenable to treatment with combined modality chemoradiation (advanced) or Stage IV (metastatic) NSCLC
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Measurable disease
* Adequate recovery from most recent systemic or local treatment for cancer
* Adequate organ function
* Life expectancy greater than or equal to (>/=) 12 weeks
* For female participants of childbearing potential and male participants, willingness to use acceptable methods of contraception

Exclusion Criteria:

* Inability to swallow oral medication
* Women who are pregnant or lactating
* Symptomatic, untreated CNS metastases
* History of malignancy other than NSCLC within 5 years prior to screening with the exception of malignancies with negligible risk of metastasis or death
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to randomization, unstable arrhythmias, or unstable angina
* Known active or uncontrolled human immunodeficiency virus (HIV) infection
* Either a concurrent condition or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or confounds the ability to interpret data from the study
* Inability to comply with other requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Percentage of Participants with Confirmed Objective Response as Assessed by the Investigator Based on the Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort B: Percentage of Participants with Confirmed Objective Response as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort C: Progression Free Survival (PFS) as Assessed by the Investigator Based on RECIST v1.1 in bTMB PP1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort D: Percentage of Participants with Confirmed Objective Response as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort E: Time in Response (TIR) as Assessed by the Investigator Based on RECIST v1.1 | Month 12
Cohort F: Investigator-Assessed Objective Response Rate (ORR) Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort G: Incidence of Adverse Events (AEs) | Baseline to last dose of study treatment + 30 days or until initiation of new anticancer therapy, whichever occurs first (up to approximately 6 years)

SECONDARY OUTCOMES:
Cohorts A-F: Duration of Response (DOR) as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A, B and D: Percentage of Participants with Clinical Benefit Response as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A, B, D, F: PFS as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A-F: Duration of Response as Assessed by the Independent Review Facility (IRF) Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A, B and D: Percentage of Participants with Clinical Benefit Response as Assessed by IRF Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A-F: PFS as Assessed by IRF Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A-F: Percentage of Participants with Confirmed Objective Response as Assessed by IRF Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohorts A-F: Overall Survival (OS) | Baseline up to approximately 6 years
Cohorts A-F: Percentage of Participants with Adverse Events (AEs) | Baseline up to approximately 6 years
Cohorts A, B, D, E, F: Percentage of Participants with Improvement Compared with Baseline in Total Severity Symptom Score as Measured by Symptoms in Lung Cancer (SILC) Scale in Patient-Reported Lung Cancer Symptoms (Cough, Dyspnea and Chest Pain) | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A-F: Time to Deterioration in Patient-Reported Lung Cancer Symptoms (Cough, Dyspnea and Chest Pain) as Measured by the SILC Scale | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts C, E, F: Change from Baseline in Patient-Reported Lung Cancer Symptom (Cough, Dyspnea, Chest pain) Score as Measured by the SILC Scale | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A-F: Change from Baseline in Health Related Quality of Life (HRQoL) Scores as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - C30 (EORTC QLQ-C30) | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A, B, D, E, F: Change from Baseline in HRQoL Scores as Measured by the SILC Scale | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A-F: Change from Baseline in Patient Functioning and Symptoms Score as Measured by the EORTC QLQ-C30 | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A, B, D, E, F: Change from Baseline in Patient Functioning and Symptoms Score as Measured by the SILC Scale | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohorts A-F: Health Status Assessed as an Index Score Using the European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | Baseline, every 4 weeks through Cycle 6 (1 Cycle = 21 or 28 days), every 8 weeks thereafter up to approximately 6 years
Cohort B: Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 to Day 28 of Cycle 1 (cycle length = 28 days)
Cohort B: Maximum Plasma Concentration (Cmax) of Alectinib | DFP: pre-dose (0 hours [hr]) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
  DFP: Dose-Finding Phase; DEP: Dose-Expanding Phase.
Cohort B: Area Under the Concentration-Time Curve from Time Zero to the Last Measurable Concentration (AUC0-last) of Alectinib | DFP: pre-dose (0 hr) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
Cohort B: Time to Reach Cmax (Tmax) of Alectinib | DFP: pre-dose (0 hr) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
Cohort B: Half-Life (t1/2) of Alectinib | DFP: pre-dose (0 hr) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
Cohort B: Metabolite to Parent Exposure Ratio for AUC0-last | DFP: pre-dose (0 hr) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
Cohort B: Metabolite to Parent Exposure Ratio for Cmax | DFP: pre-dose (0 hr) on Day 1 of Cycle 2; 0.5, 1, 2, 4, 6, 8 and 10 hr post-dose on Day 1 of Cycle 2 (1 Cycle=28 days)
Cohort C: Percentage of Participants with Objective Response as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort C: Percentage of Participants Free from Disease Progression as Assessed by the Investigator Based on RECIST v1.1 at Months 6 and 12 | Months 6, 12
Cohort C: PFS as Assessed by the Investigator based on RECIST v1.1 in bTMB PP2 | Baseline up to disease progression or death (up to approximately 6 years)
Cohort C: OS in bTMB PP2 | Baseline up to approximately 6 years
Cohort D: Time to CNS progression as Assessed by the Investigator Based on RECIST v1.1 | Baseline up to CNS progression (up to approximately 6 years)
Cohort D: Time to CNS progression as Assessed by the IRF Based on RECIST v1.1 | Baseline up to CNS progression (up to approximately 6 years)
Cohort D: Percentage of Participants who have shown improvement compared with Baseline in patient-reported cognitive function, fatigue, HRQoL, headache and vision disorder per the EORTC QLQ-C30 | Baseline, every 4 weeks until disease progression, up to approximately 6 years
Cohort D: Percentage of Participants who have shown improvement compared with Baseline in patient-reported cognitive function, fatigue, HRQoL, headache and vision disorder per the EORTC QLQ-BN20 | Baseline, every 4 weeks until disease progression, up to approximately 6 years
Cohort D: Mean Plasma Concentration of Entrectinib | Pre-dose (0 hr), 1.5 and 4 hr post-dose on Day 1 of Cycles 1, 2, 3, 4 and 5; and pre-dose on Day 1 of each subsequent treatment cycle (1 cycle = 28 days).
Cohort D: Mean Plasma Concentration of Entrectinib Metabolite M5 | Pre-dose (0 hr), 1.5 and 4 hr post-dose on Day 1 of Cycles 1, 2, 3, 4 and 5; and pre-dose on Day 1 of each subsequent treatment cycle (1 cycle = 28 days).
Cohort E: TIR as Assessed by the Investigator Based on RECIST v1.1 | Month 9
Cohort E: TIR as Assessed by IRF | Month 12
Cohorts E, F: Serum Concentration of Atezolizumab | Pre-dose (0 hr), 1.5 and 4 hr post-dose on Day 1 of Cycles 1, 2, 3, 4 and 5; and pre-dose on Day 1 of each subsequent treatment cycle (1 cycle = 28 days)
Cohorts E, F: Change from Baseline in Anti-Drug Antibodies (ADAs) | Baseline up to approximately 6 years
Cohorts E, F: Time to Confirmed Deterioration (TTCD) in Participant-Reported Lung Cancer Symptoms of Cough, Dyspnea, and Chest Pain, as Measured by the Symptoms in Lung Cancer (SILC) | Baseline up to approximately 6 years
Cohorts E, F: Proportion of Participants who Improve Compared with Baseline in Participant-Reported Lung Cancer Symptoms of Cough, Dyspnea, and Chest Pain, as Measured by the SILC | Baseline up to approximately 6 years
Cohort G: Plasma Concentration of Divarasib | Baseline up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (162):
- United States (12):
  - UC Davis, Sacramento, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - University of Kentucky, Lexington, Kentucky
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon HSU, Portland, Oregon
  - St. Luke's University Health network, Bethlehem, Pennsylvania
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
- Belgium (3):
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (4):
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System Brampton Civic Hospital, Brampton, Ontario
  - London Health Sciences Centre · Victoria Hospital, London, Ontario
  - Lakeridge Health Center, Oshawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - IUCPQ (Hôpital Laval), Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Bradford Hill Centro de Investigaciones Clinicas, Recoleta, Chile
- China (13):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - The second Xiangya hospital of central south university, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital - Sichuan University, Chengdu
  - The First Affiliated Hospital of Guangzhou Medical University Pharmacy, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Fudan Unviversity Shanghai Cancer Center, Shanghai
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- France (7):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - CHU Poitiers, Poitiers
  - Hopital Pontchaillou, Rennes
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Asklepios-Fachklinik Muenchen-Gauting, Gauting
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - HSK Dr.-Horst-Schmidt-Kliniken Klinik für Innere Medizin III Onkologie Hämatologie und Palliativmed, Wiesbaden
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hosp, Shatin
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky / Ichilov Hospital; Dept. of Oncology, Tel Aviv
- Italy (9):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO), Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST di Cremona - Azienda Socio Sanitaria Territoriale di Cremona, Cremona, Lombardy
  - Irccs Istituto Europeo di Oncologia (IEO), Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano (TO), Piedmont
- Japan (22):
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyō City
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Kanazawa University Hospital, Ishikawa
  - Kanagawa Cancer Center, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Shikoku Cancer Center, Matsuyama
  - Tohoku University Hospital, Miyagi
  - Sendai Kousei Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital, Osaka
  - Saga University Hospital, Saga
  - Shizuoka Cancer Center, Shizuoka
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Kyorin University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake-shi
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Yamaguchi - Ube Medical Center, Yamaguchi
- Mexico (4):
  - Hospital Angeles Tijuana, Tijuana, Estado de Baja California
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
- Auckland City Hospital, Auckland, New Zealand
- Hemato Oncología de Panamá Especializada, Panama City, Panama
- Peru (4):
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Instituto Peruano de Oncología y Radioterapia, Lima
  - Clinica Ricardo Palma, San Isidro
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw.Jana Pawla II, Krakow
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Centrum Onkologii Instytut im.Marii Sklodowskiej-Curie, Warsaw
- Russia (4):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow, Moscow Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Clinical Oncology Dispensary, Omsk
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - Clinical Center Nis, Niš
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (5):
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
- Spain (16):
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital General Univ. de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - ICO Badalona - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Quiron de Madrid, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan Uni Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Prince of Songkla University, Hat Yai
- Turkey (Türkiye) (7):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Medipol University Medical Faculty; Oncology Department, Istanbul
  - Marmara University Pendik Training and Research Hospital; Medikal Onkoloji, Istanbul
  - Medikal Park Izmir Hospital, Kar??yaka
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Peters S, Gadgeel SM, Mok T, Nadal E, Kilickap S, Swalduz A, Cadranel J, Sugawara S, Chiu CH, Yu CJ, Moskovitz M, Tanaka T, Nersesian R, Shagan SM, Maclennan M, Mathisen M, Bhagawati-Prasad V, Diarra C, Assaf ZJ, Archer V, Dziadziuszko R. Entrectinib in ROS1-positive advanced non-small cell lung cancer: the phase 2/3 BFAST trial. Nat Med. 2024 Jul;30(7):1923-1932. doi: 10.1038/s41591-024-03008-4. Epub 2024 Jun 19. PMID 38898120
- [Derived] Wang HY, Ho CC, Lin YT, Liao WY, Chen CY, Shih JY, Yu CJ. Comprehensive Genomic Analysis of Patients With Non-Small-Cell Lung Cancer Using Blood-Based Circulating Tumor DNA Assay: Findings From the BFAST Database of a Single Center in Taiwan. JCO Precis Oncol. 2024 Jan;8:e2300314. doi: 10.1200/PO.23.00314. PMID 38190582
- [Derived] Peters S, Dziadziuszko R, Morabito A, Felip E, Gadgeel SM, Cheema P, Cobo M, Andric Z, Barrios CH, Yamaguchi M, Dansin E, Danchaivijitr P, Johnson M, Novello S, Mathisen MS, Shagan SM, Schleifman E, Wang J, Yan M, Mocci S, Voong D, Fabrizio DA, Shames DS, Riehl T, Gandara DR, Mok T. Atezolizumab versus chemotherapy in advanced or metastatic NSCLC with high blood-based tumor mutational burden: primary analysis of BFAST cohort C randomized phase 3 trial. Nat Med. 2022 Sep;28(9):1831-1839. doi: 10.1038/s41591-022-01933-w. Epub 2022 Aug 22. PMID 35995953